CLINICAL TRIAL: NCT01425281
Title: ABSORB II RANDOMIZED CONTROLLED TRIAL A Clinical Evaluation to Compare the Safety, Efficacy and Performance of ABSORB Everolimus Eluting Bioresorbable Vascular Scaffold System Against XIENCE Everolimus Eluting Coronary Stent System in the Treatment of Subjects With Ischemic Heart Disease Caused by de Novo Native Coronary Artery Lesions
Brief Title: ABSORB II Randomized Controlled Trial
Acronym: ABSORB II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-393; CIV-11-10-002627 (Other: EUDAMED)
Record Dates: First submitted 2011-08-25; First posted 2011-08-30 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease
Keywords: Bioabsorbable; Coronary scaffold; Coronary Stent; Everolimus; Drug eluting stents; Angioplasty; Coronary artery disease; Total coronary occlusion; Coronary artery restenosis; Stent thrombosis; Myocardial ischemia; Coronary artery stenosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis; Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XIENCE™ (Active Comparator): Abbott Vascular XIENCE Everolimus Eluting Coronary Stent System
  Interventions: Device: Abbott Vascular XIENCE Everolimus Eluting Coronary Stent System
- ABSORB BVS™ (Experimental): Experimental: Abbott Vascular ABSORB Everolimus Eluting Bioresorbable Vascular Scaffold System
  Interventions: Device: Abbott Vascular ABSORB Everolimus Eluting Bioresorbable Vascular Scaffold System

INTERVENTIONS:
Device: Abbott Vascular XIENCE Everolimus Eluting Coronary Stent System — XIENCE implantation in the treatment of coronary artery disease.
  Arms: XIENCE™
Device: Abbott Vascular ABSORB Everolimus Eluting Bioresorbable Vascular Scaffold System — ABSORB BVS implantation in the treatment of coronary artery disease.
  Arms: ABSORB BVS™

SUMMARY:
Prospective, randomized (2:1), active control, single blinded, parallel two-arm, multi-center clinical investigation using Abbott Vascular ABSORB Everolimus Eluting Bioresorbable Vascular Scaffold System (ABSORB BVS); compared to Abbott Vascular XIENCE Everolimus Eluting Coronary Stent System (XIENCE)

DETAILED DESCRIPTION:
In the USA, ABSORB BVS is currently in development at Abbott Vascular. Not available for sale in the US.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

* Subject must be at least 18 years of age and less than 85 years of age.
* Subject must agree not to participate in any other clinical investigation for a period of three years following the index procedure. This includes clinical trials of medication and invasive procedures. Questionnaire-based studies, or other studies that are non-invasive and do not require medication are allowed.
* Subject is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the ABSORB BVS system and he/she or his/her legally authorized representative provides written informed consent prior to any Clinical Investigation related procedure, as approved by the appropriate Ethics Committee.
* Subject must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia).
* Subject must be an acceptable candidate for coronary artery bypass graft (CABG) surgery
* Subject must agree to undergo all clinical investigation plan-required follow-up visits, exercise testing, blood draw as well as adherence to European Society of Cardiology Guidelines and completion of quality of life questionnaires and of a subject diary to collect information including but not limited to tobacco usage, food intake, daily exercise and body weight

Angiographic Inclusion Criteria

* One or two de novo native lesions each located in a different epicardial vessel.
* If two treatable lesions meet the eligibility criteria, they must be in separate major epicardial vessels (left anterior descending (LAD) with septal and diagonal branches, left circumflex artery (LCX) with obtuse marginal and/or ramus intermedius branches and right coronary artery (RCA) and any of its branches).
* Lesion(s) must have a visually estimated diameter stenosis of ≥50% and <100% with a TIMI flow of ≥1.
* Lesion(s) must be located in a native coronary artery with Dmax by on-line quantitative coronary angiography (QCA) of ≥2.25 mm and ≤3.8 mm.
* Lesion(s) must be located in a native coronary artery with lesion(s) length by on-line QCA of ≤48 mm.
* Percutaneous interventions for lesions in a non-target vessel are allowed if done ≥30 days prior to or if planned to be done 2 years after the index procedure.
* Percutaneous intervention for lesions in the target vessel are allowed if done >6 months prior to or if planned to be done 2 years after the index procedure.

Exclusion Criteria:

* Known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, antiplatelet medication specified for use in the study (clopidogrel and prasugrel and ticlopidine, inclusive), everolimus, poly (L-lactide), poly (DL-lactide), cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated.
* Subject has a known diagnosis of acute myocardial infarction (AMI) at any time preceding the index procedure and relevant cardiac enzymes (according to local standard hospital practice) have not returned within normal limits at the time of procedure.
* Evidence of ongoing acute myocardial infarction in ECG prior to procedure
* Subject has current unstable arrhythmias.
* Left ventricular ejection fraction (LVEF) < 30%.
* Subject has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant.
* Subject is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after the procedure.
* Subject is receiving immunosuppressant therapy and/or has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus, rheumatoid arthritis, severe asthma requiring immunosuppressive medication, etc.).
* Subject is receiving chronic anticoagulation therapy that can not be stopped and restarted according to local hospital standard procedures.
* Elective surgery is planned within 2 years after the procedure that will require discontinuing either aspirin, clopidogrel, prasugrel or ticlopidine.
* Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3, a white blood cell count of <3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis)
* Known renal insufficiency (e.g., estimated glomerular filtration rate <60 ml/kg/1.73m² or serum creatinine level of >2.5 mg/dL, or subject on dialysis).
* History of bleeding diathesis or coagulopathy or will refuse blood transfusions.
* Subject has had a cerebrovascular accident (CVA) or transient ischemic neurological attack (TIA) within the past 6 months.
* Pregnant or nursing subjects and those who plan pregnancy in the period up to 3 years following index procedure. (Female subjects of child-bearing potential must have a negative pregnancy test done within 28 days prior to the index procedure and contraception must be used during participation in this trial)
* Other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) as per physician judgment that may cause non-compliance with the protocol or confound the data interpretation or is associated with a limited life expectancy.
* Subject is already participating in another clinical investigation that has not yet reached its primary endpoint.
* Subject is belonging to a vulnerable population (per investigator's judgment, e.g., subordinate hospital staff or sponsor staff) or subject unable to read or write.

Angiographic Exclusion Criteria

* Target lesion which prevents adequate (residual stenosis at target lesion(s) is ≤ 40% by visual assessment) coronary pre-dilatation.
* Target lesion in left main trunk.
* Aorto-ostial target lesion (within 3 mm of the aorta junction).
* Target lesion located within 2 mm of the origin of the LAD or LCX.
* Target lesion located distal to a diseased (vessel irregularity per angiogram and >20% stenosed lesion) arterial or saphenous vein graft.
* Target lesion involving a bifurcation lesion with side branch ≥2 mm in diameter, or with a side branch <2mm in diameter requiring guide wire protection or dilatation.
* Total occlusion (TIMI flow 0), prior to wire crossing
* Excessive tortuosity (≥ two 45° angles), or extreme angulation (≥90 °) proximal to or within the target lesion.
* Restenotic from previous intervention
* Heavy calcification proximal to or within the target lesion.
* Target lesion involves myocardial bridge.
* Target vessel contains thrombus as indicated in the angiographic images.
* Additionally clinically significant lesion(s) (≥ 40% diameter stenosis by visual assessment) for which percutaneous coronary intervention may be required <2 years after the index procedure.
* Subject has received brachytherapy in any epicardial vessel (including side branches)
* Subject has a high probability that a procedure other than pre-dilatation and study device implantation and (if necessary) post-dilatation will be required at the time of index procedure for treatment of the target vessel (e.g. atherectomy, cutting balloon)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2011-11; Primary Completion 2016-07 (Actual); Study Completion 2018-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W. Serruys, MD, PhD, Principal Investigator — Erasmus Medical Center; Bernard Chevalier, MD, Principal Investigator — Institut Jacques Cartier (ICPS)
Locations (1):
- Abbott Vascular International BVBA, Brussels, Belgium

REFERENCES:
- [Derived] Stone GW, Kimura T, Gao R, Kereiakes DJ, Ellis SG, Onuma Y, Chevalier B, Simonton C, Dressler O, Crowley A, Ali ZA, Serruys PW. Time-Varying Outcomes With the Absorb Bioresorbable Vascular Scaffold During 5-Year Follow-up: A Systematic Meta-analysis and Individual Patient Data Pooled Study. JAMA Cardiol. 2019 Dec 1;4(12):1261-1269. doi: 10.1001/jamacardio.2019.4101. PMID 31561250
- [Derived] Grundeken MJ, White RM, Hernandez JB, Dudek D, Cequier A, Haude M, van Boven AJ, Piek JJ, Helqvist S, Sabate M, Baumbach A, Suwannasom P, Ishibashi Y, Staehr P, Veldhof S, Cheong WF, de Winter RJ, Garcia-Garcia HM, Wykrzykowska JJ, Onuma Y, Serruys PW, Chevalier B. The incidence and relevance of site-reported vs. patient-reported angina: insights from the ABSORB II randomized trial comparing Absorb everolimus-eluting bioresorbable scaffold with XIENCE everolimus-eluting metallic stent. Eur Heart J Qual Care Clin Outcomes. 2016 Apr 1;2(2):108-116. doi: 10.1093/ehjqcco/qcv022. PMID 29474621
- [Derived] Ali ZA, Gao R, Kimura T, Onuma Y, Kereiakes DJ, Ellis SG, Chevalier B, Vu MT, Zhang Z, Simonton CA, Serruys PW, Stone GW. Three-Year Outcomes With the Absorb Bioresorbable Scaffold: Individual-Patient-Data Meta-Analysis From the ABSORB Randomized Trials. Circulation. 2018 Jan 30;137(5):464-479. doi: 10.1161/CIRCULATIONAHA.117.031843. Epub 2017 Oct 31. PMID 29089314
- [Derived] Serruys PW, Katagiri Y, Sotomi Y, Zeng Y, Chevalier B, van der Schaaf RJ, Baumbach A, Smits P, van Mieghem NM, Bartorelli A, Barragan P, Gershlick A, Kornowski R, Macaya C, Ormiston J, Hill J, Lang IM, Egred M, Fajadet J, Lesiak M, Windecker S, Byrne RA, Raber L, van Geuns RJ, Mintz GS, Onuma Y. Arterial Remodeling After Bioresorbable Scaffolds and Metallic Stents. J Am Coll Cardiol. 2017 Jul 4;70(1):60-74. doi: 10.1016/j.jacc.2017.05.028. PMID 28662808
- [Derived] Serruys PW, Chevalier B, Sotomi Y, Cequier A, Carrie D, Piek JJ, Van Boven AJ, Dominici M, Dudek D, McClean D, Helqvist S, Haude M, Reith S, de Sousa Almeida M, Campo G, Iniguez A, Sabate M, Windecker S, Onuma Y. Comparison of an everolimus-eluting bioresorbable scaffold with an everolimus-eluting metallic stent for the treatment of coronary artery stenosis (ABSORB II): a 3 year, randomised, controlled, single-blind, multicentre clinical trial. Lancet. 2016 Nov 19;388(10059):2479-2491. doi: 10.1016/S0140-6736(16)32050-5. Epub 2016 Oct 30. PMID 27806897
- [Derived] Sotomi Y, Ishibashi Y, Suwannasom P, Nakatani S, Cho YK, Grundeken MJ, Zeng Y, Tateishi H, Smits PC, Barragan P, Kornowski R, Gershlick AH, Windecker S, van Geuns RJ, Bartorelli AL, de Winter RJ, Tijssen J, Serruys PW, Onuma Y. Acute Gain in Minimal Lumen Area Following Implantation of Everolimus-Eluting ABSORB Biodegradable Vascular Scaffolds or Xience Metallic Stents: Intravascular Ultrasound Assessment From the ABSORB II Trial. JACC Cardiovasc Interv. 2016 Jun 27;9(12):1216-1227. doi: 10.1016/j.jcin.2016.03.022. Epub 2016 Jun 20. PMID 27339838
- [Derived] Suwannasom P, Sotomi Y, Ishibashi Y, Cavalcante R, Albuquerque FN, Macaya C, Ormiston JA, Hill J, Lang IM, Egred M, Fajadet J, Lesiak M, Tijssen JG, Wykrzykowska JJ, de Winter RJ, Chevalier B, Serruys PW, Onuma Y. The Impact of Post-Procedural Asymmetry, Expansion, and Eccentricity of Bioresorbable Everolimus-Eluting Scaffold and Metallic Everolimus-Eluting Stent on Clinical Outcomes in the ABSORB II Trial. JACC Cardiovasc Interv. 2016 Jun 27;9(12):1231-1242. doi: 10.1016/j.jcin.2016.03.027. Epub 2016 Jun 1. PMID 27262861
- [Derived] Stone GW, Gao R, Kimura T, Kereiakes DJ, Ellis SG, Onuma Y, Cheong WF, Jones-McMeans J, Su X, Zhang Z, Serruys PW. 1-year outcomes with the Absorb bioresorbable scaffold in patients with coronary artery disease: a patient-level, pooled meta-analysis. Lancet. 2016 Mar 26;387(10025):1277-89. doi: 10.1016/S0140-6736(15)01039-9. Epub 2016 Jan 27. PMID 26825231
- [Derived] Ishibashi Y, Nakatani S, Sotomi Y, Suwannasom P, Grundeken MJ, Garcia-Garcia HM, Bartorelli AL, Whitbourn R, Chevalier B, Abizaid A, Ormiston JA, Rapoza RJ, Veldhof S, Onuma Y, Serruys PW. Relation Between Bioresorbable Scaffold Sizing Using QCA-Dmax and Clinical Outcomes at 1 Year in 1,232 Patients From 3 Study Cohorts (ABSORB Cohort B, ABSORB EXTEND, and ABSORB II). JACC Cardiovasc Interv. 2015 Nov;8(13):1715-26. doi: 10.1016/j.jcin.2015.07.026. PMID 26585622
- [Derived] Ishibashi Y, Muramatsu T, Nakatani S, Sotomi Y, Suwannasom P, Grundeken MJ, Cho YK, Garcia-Garcia HM, van Boven AJ, Piek JJ, Sabate M, Helqvist S, Baumbach A, McClean D, de Sousa Almeida M, Wasungu L, Miquel-Hebert K, Dudek D, Chevalier B, Onuma Y, Serruys PW. Incidence and Potential Mechanism(s) of Post-Procedural Rise of Cardiac Biomarker in Patients With Coronary Artery Narrowing After Implantation of an Everolimus-Eluting Bioresorbable Vascular Scaffold or Everolimus-Eluting Metallic Stent. JACC Cardiovasc Interv. 2015 Jul;8(8):1053-1063. doi: 10.1016/j.jcin.2015.06.001. PMID 26205444
- [Derived] Serruys PW, Chevalier B, Dudek D, Cequier A, Carrie D, Iniguez A, Dominici M, van der Schaaf RJ, Haude M, Wasungu L, Veldhof S, Peng L, Staehr P, Grundeken MJ, Ishibashi Y, Garcia-Garcia HM, Onuma Y. A bioresorbable everolimus-eluting scaffold versus a metallic everolimus-eluting stent for ischaemic heart disease caused by de-novo native coronary artery lesions (ABSORB II): an interim 1-year analysis of clinical and procedural secondary outcomes from a randomised controlled trial. Lancet. 2015 Jan 3;385(9962):43-54. doi: 10.1016/S0140-6736(14)61455-0. Epub 2014 Sep 14. PMID 25230593
- [Derived] Diletti R, Serruys PW, Farooq V, Sudhir K, Dorange C, Miquel-Hebert K, Veldhof S, Rapoza R, Onuma Y, Garcia-Garcia HM, Chevalier B. ABSORB II randomized controlled trial: a clinical evaluation to compare the safety, efficacy, and performance of the Absorb everolimus-eluting bioresorbable vascular scaffold system against the XIENCE everolimus-eluting coronary stent system in the treatment of subjects with ischemic heart disease caused by de novo native coronary artery lesions: rationale and study design. Am Heart J. 2012 Nov;164(5):654-63. doi: 10.1016/j.ahj.2012.08.010. PMID 23137495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 501 patients (335 participants in the Absorb arm and 166 subjects in the XIENCE arm) were randomized into the ABSORB II Randomized controlled trial (RCT) at 46 international outside the United States (OUS) sites study sites. First subject was randomized on 28 November 2011 and the last subject randomized on 04 June 2013.
Pre-assignment Details: Early termination by 5-year affected 120 patients due to subject withdrew consent (n=20), withdrawn by the site (n=1), lost to follow-up (n=9), death (n=20),early termination due to a lapse in the protocol renewal by the Polish Ethics Committee (n=37) and early terminations due to 'other' reasons (n=33).
Groups:
- Absorb BVS™: Abbott Vascular Absorb Everolimus Eluting Bioresorbable Vascular Scaffold System: ABSORB bioresorbable vascular scaffold (Absorb BVS) implantation in the treatment of coronary artery disease.
Period: At 30-day Clinical Follow-up
Arm/Group | Absorb BVS™ | XIENCE™
Started | 335 (Intent-to-Treat (ITT) Population) | 166 (Intent-to-Treat (ITT) Population)
Completed | 334 | 166
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: At 180-day Clinical Follow-up
Arm/Group | Absorb BVS™ | XIENCE™
Started | 334 | 166
Completed | 331 | 165
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Death | 0 | 1
Period: At 1-year Clinical Follow-up
Arm/Group | Absorb BVS™ | XIENCE™
Started | 331 | 165
Completed | 329 | 164
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Withdrawal by Physician/Site | 1 | 0
Period: At 2-year Clinical Follow-up
Arm/Group | Absorb BVS™ | XIENCE™
Started | 329 | 164
Completed | 323 | 163
Not Completed | 6 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Patient did not want to participate in t | 1 | 0
Period: At 3-year Clinical Follow-up
Arm/Group | Absorb BVS™ | XIENCE™
Started | 323 | 163
Completed | 318 | 157
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Death | 2 | 3
Period: At 4-year Clinical Follow-up
Arm/Group | Absorb BVS™ | XIENCE™
Started | 318 | 157
Completed | 288 | 136
Not Completed | 30 | 21
Not completed — Death | 7 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Did not consent for follow-up after 3 ye | 10 | 10
Not completed — Terminated by Polish Ethics Committee | 6 | 5
Not completed — Lost to Follow-up | 4 | 1
Period: At 5-year Clinical Follow-up
Arm/Group | Absorb BVS™ | XIENCE™
Started | 288 | 136
Completed | 256 | 125
Not Completed | 32 | 11
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Terminated by Polish Ethics Committee | 19 | 7
Not completed — Refused/terminated | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Absorb BVS™ | XIENCE™ | Total
Number analyzed (Participants) | 335 | 166 | 501
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 202 | 102 | 304
  >=65 years | 133 | 64 | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (10.0) | 60.9 (10.0) | 61.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 34 | 116
  Male | 253 | 132 | 385
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 4 | 4 | 8
  Belgium | 6 | 0 | 6
  Denmark | 11 | 5 | 16
  France | 51 | 25 | 76
  Germany | 14 | 6 | 20
  Israel | 8 | 4 | 12
  Italy | 33 | 13 | 46
  Netherlands | 48 | 34 | 82
  New Zealand | 15 | 8 | 23
  Poland | 26 | 16 | 42
  Portugal | 11 | 2 | 13
  Spain | 63 | 28 | 91
  Switzerland | 8 | 4 | 12
  United Kingdom | 37 | 17 | 54

OUTCOME MEASURES:

1. Primary Outcome: Absolute Difference (3 Years Post Nitrate- 3 Years Pre Nitrate) In-Scaffold Mean Lumen Diameter (MLD)
Description: In-scaffold:Within the margins of the scaffold.
Time Frame: 3 years
Population: ITT population. The number of participants analyzed includes subjects who had available follow up data at that time frame
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 239 | 121
Number analyzed (Target lesions) | 258 | 130
mm | 0.05 (0.11) | 0.06 (0.12)
Statistical Analysis 1: Comparison: Absorb BVS™ vs XIENCE™; Angiographic vasomotion reactivity following nitrate administration, the test was analyzable for 388 paired lesions (Absorb arm [258 lesions] vs Xience arm [130 lesions]); Test type: Superiority; p = 0.49, t-test, 2 sided; Null and alternative hypotheses for superiority testing. H0: EndpointABSORB BVS = EndpointXIENCE H1: EndpointABSORB BVS ≠ EndpointXIENCE

2. Primary Outcome: Absolute Difference (3 Years Post-nitrate - Post Procedure Post-nitrate) In-Scaffold Minimum Lumen Diameter
Description: In-scaffold:Within the margins of the scaffold.
Time Frame: 3 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 275 | 138
Number analyzed (Target lesions) | 298 | 151
mm | -0.37 (0.45) | -0.25 (0.25)
Statistical Analysis 1: Comparison: Absorb BVS™ vs XIENCE™; Follow-up angiographic analysis was available for 298 lesions in the Absorb arm and 151 lesions in the Xience arm; Test type: Non-Inferiority — Using t-test with non-inferiority margin of 0.140mm; p = 0.78, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Device Success
Description: Successful delivery and deployment of the first study scaffold/stent the intended target lesion and successful withdrawal of the delivery system with attainment of final in-scaffold/stent residual stenosis of less than 50% by quantitative coronary angiography (QCA).
Time Frame: From the start of index procedure to end of index procedure
Population: Device Success is measured on a per Lesion basis. Some patients had more than one lesion treated so the total number of lesions is larger than the number of patients.
Measure: Number; unit: Percentage of lesions
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 335 | 162
Number analyzed (Target lesions) | 364 | 182
Percentage of lesions | 99.5 | 100

4. Secondary Outcome: Number of Participants With Procedural Success
Description: Achievement of final in-scaffold/stent residual stenosis of less than 50% by QCA with successful delivery and deployment of at least one study scaffold/stent at the intended target lesion and successful withdrawal of the delivery system for all target lesions without the occurrence of cardiac death, target vessel MI or repeat TLR during the hospital stay.
Time Frame: From the start of index procedure to end of index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 335 | 166
Participants | 322 | 164

5. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in subjects with coexisting potentially fatal non-cardiac disease (e.g. cancer, infection) should be classified as cardiac.
  * Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  * Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  * Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Time Frame: In-hospital (≤ 7 days of post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 335 | 166
Participants | 0 | 0

6. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in subjects with coexisting potentially fatal non-cardiac disease (e.g. cancer, infection) should be classified as cardiac.
  • Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  • Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  • Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 334 | 166
Participants | 0 | 0

7. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 6
Time Frame: 180 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 332 | 166
Participants | 0 | 1

8. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 6
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 331 | 165
Participants | 0 | 1

9. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 6
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 327 | 164
Participants | 4 | 1

10. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 6
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 325 | 161
Participants | 8 | 6

11. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 5
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 308 | 147
Participants | 11 | 7

12. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 5
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 285 | 138
Participants | 13 | 7

13. Secondary Outcome: Number of Participants With All Myocardial Infarction (Per Protocol Definition)
Description: Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Elevation of Creatine kinase (CK) levels to ≥ two times the upper limit of normal (ULN) with elevated Creatine kinase-MB (CK-MB) in the absence of new pathological Q waves.
Time Frame: In-hospital (≤ 7 days of post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 335 | 166
Participants | 13 | 2

14. Secondary Outcome: Number of Participants With All Myocardial Infarction (Per Protocol Definition)
Description: as for outcome 13
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 334 | 166
Participants | 14 | 2

15. Secondary Outcome: Number of Participants With All Myocardial Infarction (Per Protocol Definition)
Description: Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 332 | 166
Participants | 14 | 2

16. Secondary Outcome: Number of Participants With All Myocardial Infarction (Per Protocol Definition)
Description: as for outcome 15
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 331 | 165
Participants | 15 | 2

17. Secondary Outcome: Number of Participants With All Myocardial Infarction (Per Protocol Definition)
Description: as for outcome 15
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 327 | 164
Participants | 19 | 4

18. Secondary Outcome: Number of Participants With All Myocardial Infarction (Per Protocol Definition)
Description: as for outcome 15
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 325 | 161
Participants | 27 | 5

19. Secondary Outcome: Number of Participants With All Myocardial Infarction (Per Protocol Definition)
Description: Myocardial Infarction (MI)
  * Q wave MI: Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 308 | 147
Participants | 27 | 5

20. Secondary Outcome: Number of Participants With All Myocardial Infarction (Per Protocol Definition)
Description: as for outcome 19
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 285 | 138
Participants | 27 | 6

21. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: Target Lesion Revascularization is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLR should be classified prospectively as clinically indicated (CI) or not clinically indicated by the investigator prior to repeat angiography. An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement.
  The target lesion is defined as the treated segment from 5 mm proximal to the stent and to 5 mm distal to the scaffold/stent.
Time Frame: In-hospital (≤ 7 days of post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 335 | 166
Participants | 1 | 0

22. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 21
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 334 | 166
Participants | 2 | 0

23. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: Target Lesion Revascularization is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLR should be classified prospectively as clinically indicated [CI] or not clinically indicated by the investigator prior to repeat angiography. An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement.
  The target lesion is defined as the treated segment from 5 mm proximal to the stent and to 5 mm distal to the scaffold/stent.
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 332 | 166
Participants | 2 | 1

24. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 23
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 331 | 165
Participants | 4 | 3

25. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 23
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 327 | 164
Participants | 9 | 3

26. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 23
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 325 | 161
Participants | 24 | 8

27. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 23
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 308 | 147
Participants | 27 | 8

28. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 23
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 285 | 138
Participants | 28 | 8

29. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: Target Vessel Revascularization is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion which includes upstream and downstream branches and the target lesion itself.
Time Frame: In-hospital (≤ 7 days of post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 335 | 166
Participants | 1 | 0

30. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 29
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 334 | 166
Participants | 2 | 2

31. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 29
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 332 | 166
Participants | 4 | 4

32. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 29
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 331 | 165
Participants | 8 | 8

33. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 29
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 327 | 164
Participants | 15 | 9

34. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 29
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 325 | 161
Participants | 33 | 19

35. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 29
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 308 | 147
Participants | 38 | 19

36. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 29
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 285 | 138
Participants | 41 | 19

37. Secondary Outcome: Number of Participants With Non Target Vessel Revascularization (Non-TVR)
Description: Non Target Vessel Revascularization (Non-TVR)is any revascularization in a vessel other than the target vessel.
Time Frame: In-hospital (≤ 7 days of post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 335 | 166
Participants | 0 | 0

38. Secondary Outcome: Number of Participants With Non Target Vessel Revascularization (Non-TVR)
Description: Non Target Vessel Revascularization (Non-TVR)is any revascularization in a vessel other than the target vessel.
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 334 | 166
Participants | 1 | 0

39. Secondary Outcome: Number of Participants With Non Target Vessel Revascularization (Non-TVR)
Description: Non Target Vessel Revascularization (Non-TVR)is any revascularization in a vessel other than the target vessel.
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 332 | 166
Participants | 4 | 3

40. Secondary Outcome: Number of Participants With Non Target Vessel Revascularization (Non-TVR)
Description: Non Target Vessel Revascularization (Non-TVR)is any revascularization in a vessel other than the target vessel.
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 331 | 165
Participants | 6 | 6

41. Secondary Outcome: Number of Participants With Non Target Vessel Revascularization (Non-TVR)
Description: Non Target Vessel Revascularization (Non-TVR)is any revascularization in a vessel other than the target vessel.
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 327 | 164
Participants | 10 | 11

42. Secondary Outcome: Number of Participants With Non Target Vessel Revascularization (Non-TVR)
Description: Non Target Vessel Revascularization (Non-TVR)is any revascularization in a vessel other than the target vessel.
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 325 | 161
Participants | 22 | 19

43. Secondary Outcome: Number of Participants With Non Target Vessel Revascularization (Non-TVR)
Description: Non Target Vessel Revascularization (Non-TVR)is any revascularization in a vessel other than the target vessel.
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 308 | 147
Participants | 29 | 20

44. Secondary Outcome: Number of Participants With Non-Target Vessel Revascularization (Non-TVR)
Description: Non Target Vessel Revascularization (Non-TVR) is any revascularization in a vessel other than the target vessel.
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 285 | 138
Participants | 30 | 20

45. Secondary Outcome: Number of Participants With All Revascularization
Description: Revascularization:
  Target Lesion Revascularization (TLR) is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. The target lesion is defined as the treated segment from 5 mm proximal to the scaffold and to 5 mm distal to the test scaffold.
  Target Vessel Revascularization (TVR) is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion.
  Non Target Lesion Revascularization (Non-TLR) is any revascularization in the target vessel for a lesion other than the target lesion.
  Non Target Vessel Revascularization (Non-TVR)is any revascularization in a vessel other than the target vessel.
Time Frame: In-hospital (≤ 7 days of post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 335 | 166
Participants | 1 | 0

46. Secondary Outcome: Number of Participants With All Revascularization
Description: Revascularization:
  * Target Lesion Revascularization (TLR) is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. The target lesion is defined as the treated segment from 5 mm proximal to the scaffold and to 5 mm distal to the test scaffold.
  * Target Vessel Revascularization (TVR) is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion.
  * Non Target Lesion Revascularization (Non-TLR) is any revascularization in the target vessel for a lesion other than the target lesion.
  * Non Target Vessel Revascularization (Non-TVR)is any revascularization in a vessel other than the target vessel.
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 334 | 166
Participants | 2 | 2

47. Secondary Outcome: Number of Participants With All Revascularization
Description: as for outcome 46
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 332 | 166
Participants | 7 | 6

48. Secondary Outcome: Number of Participants With All Revascularization
Description: as for outcome 46
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 331 | 165
Participants | 12 | 12

49. Secondary Outcome: Number of Participants With All Revascularization
Description: as for outcome 46
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 327 | 164
Participants | 22 | 18

50. Secondary Outcome: Number of Participants With All Revascularization
Description: as for outcome 46
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 325 | 161
Participants | 49 | 33

51. Secondary Outcome: Number of Participants With All Revascularization
Description: as for outcome 46
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 308 | 147
Participants | 57 | 34

52. Secondary Outcome: Number of Participants With All Revascularization
Description: as for outcome 45
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 285 | 138
Participants | 59 | 34

53. Secondary Outcome: Number of Participants Experiencing All Death/All MI
Description: All deaths includes
  * Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  * Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  * Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
  Myocardial Infarction (MI) Q wave MI Development of new, pathological Q wave on the ECG. Non-Q wave MI Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: In-hospital (≤ 7 days of post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 335 | 166
Participants | 13 | 2

54. Secondary Outcome: Number of Participants Experiencing All Death/All MI
Description: All deaths includes
  • Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  • Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  • Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
  Myocardial Infarction (MI)
  * Q wave MI Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 334 | 166
Participants | 14 | 2

55. Secondary Outcome: Number of Participants Experiencing All Death/All MI
Description: as for outcome 54
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 332 | 166
Participants | 14 | 3

56. Secondary Outcome: Number of Participants Experiencing All Death/All MI
Description: All deaths includes
  * Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  * Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  * Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
  Myocardial Infarction (MI)
  * Q wave MI: Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 331 | 165
Participants | 15 | 3

57. Secondary Outcome: Number of Participants Experiencing All Death/All MI
Description: All deaths includes
  * Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), un witnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  * Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  * Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
  Myocardial Infarction (MI)
  * Q wave MI: Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 327 | 164
Participants | 22 | 5

58. Secondary Outcome: Number of Participants Experiencing All Death/All MI
Description: as for outcome 57
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 325 | 161
Participants | 33 | 11

59. Secondary Outcome: Number of Participants Experiencing All Death/All MI
Description: as for outcome 57
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 308 | 147
Participants | 35 | 12

60. Secondary Outcome: Number of Participants Experiencing All Death/All MI
Description: All deaths includes
  * Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  * Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  * Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma. Myocardial Infarction (MI)
  * Q wave MI Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 285 | 138
Participants | 37 | 13

61. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF) (Cardiac Death,(Target Vessel Myocardial Infarction(TV-MI), ID-TLR)
Description: Target Lesion Failure is composite of Cardiac death/ Target Vessel Myocardial Infarction (TV-MI)/ Ischemic-Driven Target Lesion Revascularization (ID-TLR).
Time Frame: In-hospital (≤ 7 days of post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 335 | 166
Participants | 12 | 2

62. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF) (Cardiac Death, Target Vessel Myocardial Infarction (TV-MI), ID-TLR)
Description: as for outcome 61
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 334 | 166
Participants | 13 | 2

63. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF) (Cardiac Death, TV-MI, ID-TLR)
Description: as for outcome 61
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 332 | 166
Participants | 13 | 3

64. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF) (Cardiac Death, TV-MI, ID-TLR)
Description: as for outcome 61
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 331 | 165
Participants | 16 | 5

65. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF) (Cardiac Death, TV-MI, ID-TLR)
Description: as for outcome 61
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 327 | 164
Participants | 23 | 5

66. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF) (Cardiac Death, TV-MI, ID-TLR)
Description: as for outcome 61
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 325 | 161
Participants | 34 | 8

67. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF) (Cardiac Death, TV-MI, ID-TLR)
Description: as for outcome 61
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 308 | 147
Participants | 37 | 9

68. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF) (Cardiac Death, TV-MI, ID-TLR)
Description: as for outcome 61
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 285 | 138
Participants | 38 | 9

69. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE) (Cardiac Death, All MI, ID-TLR)
Description: Major adverse cardiac events (MACE) is defined as the composite of cardiac death, all myocardial infarction, and ischemic driven target lesion revascularization (ID-TLR).
Time Frame: In-hospital (≤ 7 days of post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 335 | 166
Participants | 13 | 2

70. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE) (Cardiac Death, All MI, ID-TLR)
Description: as for outcome 69
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 334 | 166
Participants | 14 | 2

71. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE) (Cardiac Death, All MI, ID-TLR)
Description: as for outcome 69
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 332 | 166
Participants | 14 | 3

72. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE) (Cardiac Death, All MI, ID-TLR)
Description: as for outcome 69
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 331 | 165
Participants | 17 | 5

73. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE) (Cardiac Death, All MI, ID-TLR)
Description: as for outcome 69
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 327 | 164
Participants | 25 | 7

74. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE) (Cardiac Death, All MI, ID-TLR)
Description: as for outcome 69
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 325 | 161
Participants | 38 | 11

75. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE) (Cardiac Death, All MI, ID-TLR)
Description: as for outcome 69
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 308 | 147
Participants | 40 | 12

76. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE) (Cardiac Death, All MI, ID-TLR)
Description: as for outcome 69
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 285 | 138
Participants | 41 | 13

77. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF) (Cardiac Death, All MI, ID-TVR)
Description: Target Vessel Failure (TVF) is the composite of Cardiac Death, Myocardial infarction (MI) or Ischemic-Driven Target Vessel Revascularization (ID-TVR).
Time Frame: In-hospital (≤ 7 days of post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 335 | 166
Participants | 13 | 2

78. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF) (Cardiac Death, All MI, ID-TVR)
Description: as for outcome 77
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 334 | 166
Participants | 14 | 3

79. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF) (Cardiac Death, All MI, ID-TVR)
Description: as for outcome 77
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 332 | 166
Participants | 15 | 5

80. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF) (Cardiac Death, All MI, ID-TVR)
Description: as for outcome 77
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 331 | 165
Participants | 18 | 8

81. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF) (Cardiac Death, All MI, ID-TVR)
Description: as for outcome 77
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 327 | 164
Participants | 28 | 11

82. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF) (Cardiac Death, All MI, ID-TVR)
Description: as for outcome 77
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 325 | 161
Participants | 41 | 20

83. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF) (Cardiac Death, All MI, ID-TVR)
Description: as for outcome 77
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 308 | 147
Participants | 45 | 21

84. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF) (Cardiac Death, All MI, ID-TVR)
Description: as for outcome 77
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 285 | 138
Participants | 47 | 22

85. Secondary Outcome: Number of Participants With DMR (All Death, All MI, All Revascularization)
Description: DMR is the composite of All Death, All MI, All Revascularization
Time Frame: In-hospital (≤ 7 days of post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 335 | 166
Participants | 13 | 2

86. Secondary Outcome: Number of Participants With DMR (All Death, All MI, All Revascularization)
Description: DMR is the composite of All Death, All MI, All Revascularization.
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 334 | 166
Participants | 14 | 4

87. Secondary Outcome: Number of Participants With DMR (All Death, All MI, All Revascularization)
Description: DMR is the composite of All Death, All MI, All Revascularization.
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 332 | 166
Participants | 19 | 9

88. Secondary Outcome: Number of Participants With DMR (All Death, All MI, All Revascularization)
Description: DMR is the composite of All Death, All MI, All Revascularization.
Time Frame: 1 year
Population: Intent-to-Treat Population (ITT).The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 331 | 165
Participants | 24 | 15

89. Secondary Outcome: Number of Participants With DMR (All Death, All MI, All Revascularization)
Description: DMR is the composite of All Death, All MI, All Revascularization.
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 327 | 164
Participants | 38 | 21

90. Secondary Outcome: Number of Participants With DMR (All Death, All MI, All Revascularization)
Description: DMR is the composite of All Death, All MI, All Revascularization.
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 325 | 161
Participants | 68 | 39

91. Secondary Outcome: Number of Participants With DMR (All Death, All MI, All Revascularization)
Description: DMR is the composite of All Death, All MI, All Revascularization
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 308 | 147
Participants | 76 | 40

92. Secondary Outcome: Number of Participants With DMR (All Death, All MI, All Revascularization)
Description: DMR is the composite of All Death, All MI, All Revascularization
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 285 | 138
Participants | 80 | 41

93. Secondary Outcome: Number of Participants Experiencing Cardiac Death/All MI
Description: Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), un witnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Myocardial Infarction (MI) Q wave MI: Development of new, pathological Q wave on the ECG. Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves
Time Frame: In-hospital (≤ 7 days of post index procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 335 | 166
Participants | 13 | 2

94. Secondary Outcome: Number of Participants Experiencing Cardiac Death/All MI
Description: Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), un witnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Myocardial Infarction (MI)
  * Q wave MI: Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 334 | 166
Participants | 14 | 2

95. Secondary Outcome: Number of Participants Experiencing Cardiac Death/All MI
Description: as for outcome 94
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 332 | 166
Participants | 14 | 2

96. Secondary Outcome: Number of Participants Experiencing Cardiac Death/All MI
Description: as for outcome 94
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 331 | 165
Participants | 15 | 2

97. Secondary Outcome: Number of Participants Experiencing Cardiac Death/All MI
Description: as for outcome 94
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 327 | 164
Participants | 20 | 4

98. Secondary Outcome: Number of Participants Experiencing Cardiac Death/All MI
Description: as for outcome 94
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 325 | 161
Participants | 28 | 8

99. Secondary Outcome: Number of Participants Experiencing Cardiac Death/All MI
Description: as for outcome 93
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 308 | 147
Participants | 29 | 9

100. Secondary Outcome: Number of Participants Experiencing Cardiac Death/All MI
Description: as for outcome 93
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 285 | 138
Participants | 29 | 10

101. Secondary Outcome: Number of Participants With Acute Stent/Scaffold Thrombosis
Description: Scaffold/Stent thrombosis should be reported as a cumulative value at the different time points.
  Timings:
  Acute:0-24 hours;Subacute:>24 hours-30 days;Late:30 days-1 year;Very late:>1 year.
  Definite stent thrombosis occurred by either angiographic/pathologic confirmation.
  Angiographic confirmation:The presence of a thrombus that originates in the stent or in the segment 5 mm proximal or distal to the stent&presence of at least 1 of the following criteria within a 48-hour time window
  -Acute onset of ischemic symptoms at rest;New ischemic ECG changes;Typical rise&fall in cardiac biomarkers;Nonocclusive/Occlusive thrombus
  Pathological confirmation:Evidence of recent thrombus.
  Probable stent thrombosis may occur after intracoronary stenting due to:
  * Unexplained death within first 30 days
  * Any MI that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis&in the absence of any other obvious cause.
Time Frame: <=1 day
Population: ITT population. .
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 335 | 166
Participants
  Definite | 1 | 0
  Probable | 0 | 0

102. Secondary Outcome: Number of Participants With Subacute Stent/Scaffold Thrombosis
Description: as for outcome 101
Time Frame: > 1-30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 334 | 166
Participants
  Definite | 1 | 0
  Probable | 0 | 0

103. Secondary Outcome: Number of Participants With Acute/Subacute Stent/Scaffold Thrombosis
Description: as for outcome 101
Time Frame: 0-30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 334 | 166
Participants
  Definite | 2 | 0
  Probable | 0 | 0

104. Secondary Outcome: Number of Participants With Late Stent/Scaffold Thrombosis
Description: as for outcome 101
Time Frame: 31-365 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 329 | 164
Participants
  Definite | 0 | 0
  Probable | 1 | 0

105. Secondary Outcome: Number of Participants With Very Late Stent/Scaffold Thrombosis
Description: as for outcome 101
Time Frame: > 365 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 329 | 164
Participants
  Definite | 6 | 0
  Probable | 0 | 0

106. Secondary Outcome: Number of Participants With Cumulative Stent/Scaffold Thrombosis
Description: as for outcome 101
Time Frame: 0-1853 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS™ | XIENCE™
Number analyzed (Participants) | 263 | 129
Participants
  Definite | 8 | 0
  Probable | 1 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | XIENCE™ | Absorb BVS™
All-Cause Mortality (participants affected / at risk) | 7/138 | 13/285
Serious Adverse Events (participants affected / at risk) | 84/159 | 165/318
Other Adverse Events (participants affected / at risk) | 151/159 | 296/318
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XIENCE™ (N=159) | Absorb BVS™ (N=318)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 11
ANGINA PECTORIS (Cardiac disorders) | 27 | 42
ANGINA UNSTABLE (Cardiac disorders) | 4 | 5
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 7
ATRIAL FLUTTER (Cardiac disorders) | 1 | 2
ATRIAL TACHYCARDIA (Cardiac disorders) | 1 | 0
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1 | 1
BUNDLE BRANCH BLOCK (Cardiac disorders) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 0 | 2
CARDIAC FAILURE (Cardiac disorders) | 0 | 2
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 3
CORONARY ARTERY DISSECTION (Cardiac disorders) | 2 | 3
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 2 | 0
CORONARY ARTERY PERFORATION (Cardiac disorders) | 0 | 2
CORONARY ARTERY STENOSIS (Cardiac disorders) | 5 | 5
CORONARY ARTERY THROMBOSIS (Cardiac disorders) | 0 | 3
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 4 | 5
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 2 | 4
PALPITATIONS (Cardiac disorders) | 1 | 1
PERICARDITIS (Cardiac disorders) | 1 | 0
SICK SINUS SYNDROME (Cardiac disorders) | 0 | 2
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 2
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 0 | 1
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 | 2
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | 2
BICUSPID AORTIC VALVE (Congenital, familial and genetic disorders) | 0 | 1
HYDROCELE (Congenital, familial and genetic disorders) | 0 | 1
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 0 | 1
CATARACT (Eye disorders) | 0 | 4
MACULAR DEGENERATION (Eye disorders) | 0 | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 2
ENTEROCOLITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 1
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 2
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
HAEMATEMESIS (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0
MESENTERIC ARTERY STENOSIS (Gastrointestinal disorders) | 0 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1
ADVERSE DRUG REACTION (General disorders) | 0 | 1
CATHETER SITE HAEMATOMA (General disorders) | 0 | 1
CATHETER SITE HAEMORRHAGE (General disorders) | 0 | 1
CHEST DISCOMFORT (General disorders) | 1 | 0 — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS.
CHEST PAIN (General disorders) | 3 | 4 — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS.
DEATH (General disorders) | 2 | 1 — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS.
MICROLITHIASIS (General disorders) | 1 | 0 — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS.
NON-CARDIAC CHEST PAIN (General disorders) | 3 | 11 — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS.
Other (General disorders) | 8 | 16
PELVIC MASS (General disorders) | 0 | 1
SUDDEN DEATH (General disorders) | 0 | 1
THROMBOSIS IN DEVICE (General disorders) | 0 | 3
VASCULAR COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 2
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 1 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 0 | 1
APPENDICITIS (Infections and infestations) | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 1
CYSTITIS (Infections and infestations) | 0 | 1
DOUGLAS' ABSCESS (Infections and infestations) | 1 | 0
ERYSIPELAS (Infections and infestations) | 1 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 2
GINGIVAL INFECTION (Infections and infestations) | 0 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1
OSTEOMYELITIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 3 | 5
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 | 0
UROSEPSIS (Infections and infestations) | 0 | 1
CATHETER SITE ABSCESS (Infections and infestations) | 0 | 1
ORCHITIS (Infections and infestations) | 0 | 2
PYELONEPHRITIS (Infections and infestations) | 0 | 2
SEPSIS (Infections and infestations) | 0 | 3
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
CATHETER SITE HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 0 | 2
ESCHAR (Injury, poisoning and procedural complications) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 2 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
LIMB CRUSHING INJURY (Injury, poisoning and procedural complications) | 1 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 1
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
NERVE ROOT INJURY LUMBAR (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL MYOCARDIAL INFARCTION (Injury, poisoning and procedural complications) | 1 | 2
POSTOPERATIVE FEVER (Injury, poisoning and procedural complications) | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SPINAL CORD INJURY (Injury, poisoning and procedural complications) | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 1
CONFUSION POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 | 1
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 0 | 5
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
CARDIAC STRESS TEST ABNORMAL (Investigations) | 1 | 3
ELECTROCARDIOGRAM ST SEGMENT DEPRESSION (Investigations) | 1 | 0
ELECTROCARDIOGRAM ST SEGMENT ABNORMAL (Investigations) | 0 | 1
EXERCISE TEST ABNORMAL (Investigations) | 0 | 2
BIOPSY PROSTATE (Investigations) | 0 | 1
BLOOD GLUCOSE ABNORMAL (Investigations) | 0 | 1
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 0 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1
OBESITY (Metabolism and nutrition disorders) | 1 | 1
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 | 2
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
DUPUYTREN'S CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 2
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 0 | 1
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 0 | 1
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
BENIGN SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLON NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GLIOBLASTOMA MULTIFORME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
LEUKAEMIA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SCROTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SMALL INTESTINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SMALL INTESTINE CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
GASTROINTESTINAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
GASTROOESOPHAGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 | 3
DIZZINESS (Nervous system disorders) | 1 | 0
EPILEPSY (Nervous system disorders) | 0 | 1
HYDROCEPHALUS (Nervous system disorders) | 1 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0
PRE SYNCOPE (Nervous system disorders) | 1 | 0
SENSORY LOSS (Nervous system disorders) | 2 | 0
SYNCOPE (Nervous system disorders) | 3 | 3
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
CLONIC CONVULSION (Nervous system disorders) | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 2
DEPRESSION (Psychiatric disorders) | 1 | 0
MENTAL DISORDER (Psychiatric disorders) | 0 | 3
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 0 | 1
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 1 | 0
URINARY TRACT DISORDER (Renal and urinary disorders) | 0 | 2
VESICAL FISTULA (Renal and urinary disorders) | 1 | 0
RENAL ANEURYSM (Renal and urinary disorders) | 0 | 1
CALCULUS URINARY (Renal and urinary disorders) | 0 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 2
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 4
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
SHOULDER OPERATION (Surgical and medical procedures) | 0 | 1
SPINAL LAMINECTOMY (Surgical and medical procedures) | 1 | 0
INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 1 | 0
AORTIC STENOSIS (Vascular disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 1
TEMPORAL ARTERITIS (Vascular disorders) | 0 | 1
AORTIC ANEURYSM (Vascular disorders) | 2 | 0
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 1 | 1
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 | 1
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 0 | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 1 | 1
INTERMITTENT CLAUDICATION (Vascular disorders) | 0 | 1
VARICOSE VEIN (Vascular disorders) | 0 | 1
ARRHYTHMIA (Cardiac disorders) | 0 | 1
CEREBRAL HAEMATOMA (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XIENCE™ (N=159) | Absorb BVS™ (N=318)
ANAEMIA (Blood and lymphatic system disorders) | 3 | 5
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 2
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 2
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 12
ANGINA PECTORIS (Cardiac disorders) | 54 | 87
ANGINA UNSTABLE (Cardiac disorders) | 5 | 5
ARRHYTHMIA (Cardiac disorders) | 1 | 1
ARTERIOSPASM CORONARY (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 4 | 10
ATRIAL FLUTTER (Cardiac disorders) | 1 | 2
ATRIAL TACHYCARDIA (Cardiac disorders) | 1 | 0
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1 | 1
BRADYCARDIA (Cardiac disorders) | 2 | 1
CARDIAC FAILURE (Cardiac disorders) | 0 | 6
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 3
CORONARY ARTERY DISSECTION (Cardiac disorders) | 6 | 7
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 2 | 1
CORONARY ARTERY PERFORATION (Cardiac disorders) | 0 | 2
CORONARY ARTERY STENOSIS (Cardiac disorders) | 5 | 6
CORONARY ARTERY THROMBOSIS (Cardiac disorders) | 0 | 3
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 4 | 5
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 3 | 10
PALPITATIONS (Cardiac disorders) | 3 | 5
PERICARDITIS (Cardiac disorders) | 1 | 1
PRINZMETAL ANGINA (Cardiac disorders) | 1 | 0
SICK SINUS SYNDROME (Cardiac disorders) | 0 | 2
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 3
TACHYCARDIA (Cardiac disorders) | 1 | 1
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 0 | 1
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 | 1
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 | 3
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | 5
ATRIOVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 1
BUNDLE BRANCH BLOCK (Cardiac disorders) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 0 | 2
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 1
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 1
TACHYARRHYTHMIA (Cardiac disorders) | 0 | 1
BICUSPID AORTIC VALVE (Congenital, familial and genetic disorders) | 0 | 1
HYDROCELE (Congenital, familial and genetic disorders) | 0 | 1
CERUMEN IMPACTION (Ear and labyrinth disorders) | 0 | 2
EXTERNAL EAR PAIN (Ear and labyrinth disorders) | 0 | 1
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 0 | 2
TINNITUS (Ear and labyrinth disorders) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 1 | 2
AURICULAR PERICHONDRITIS (Ear and labyrinth disorders) | 0 | 1
BASEDOW'S DISEASE (Endocrine disorders) | 1 | 0
GOITRE (Endocrine disorders) | 1 | 0
HYPOTHYROIDISM (Endocrine disorders) | 0 | 2
THYROIDITIS CHRONIC (Endocrine disorders) | 0 | 1
AGE-RELATED MACULAR DEGENERATION (Eye disorders) | 0 | 1
CATARACT (Eye disorders) | 0 | 7
CHOROIDAL HAEMORRHAGE (Eye disorders) | 0 | 1
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 | 2
CORNEAL EROSION (Eye disorders) | 0 | 1
DIABETIC RETINOPATHY (Eye disorders) | 1 | 1
EYE HAEMORRHAGE (Eye disorders) | 1 | 0
EYE PRURITUS (Eye disorders) | 0 | 1
GLAUCOMA (Eye disorders) | 0 | 1
KERATITIS (Eye disorders) | 0 | 2
MACULAR OEDEMA (Eye disorders) | 0 | 1
OCULAR DISCOMFORT (Eye disorders) | 0 | 1
ULCERATIVE KERATITIS (Eye disorders) | 0 | 1
UVEITIS (Eye disorders) | 0 | 1
VISION BLURRED (Eye disorders) | 1 | 2
VISUAL IMPAIRMENT (Eye disorders) | 0 | 1
IRIDOCYCLITIS (Eye disorders) | 0 | 1
MACULAR DEGENERATION (Eye disorders) | 0 | 1
MACULAR HOLE (Eye disorders) | 0 | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 2 | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 4
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 | 6
ANAL FISSURE (Gastrointestinal disorders) | 1 | 0
ANAL FISTULA (Gastrointestinal disorders) | 1 | 0
COLONIC POLYP (Gastrointestinal disorders) | 0 | 4
CONSTIPATION (Gastrointestinal disorders) | 1 | 3
DIARRHOEA (Gastrointestinal disorders) | 4 | 5
DIVERTICULUM (Gastrointestinal disorders) | 1 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 1
DYSPEPSIA (Gastrointestinal disorders) | 4 | 5
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1
GASTRIC DISORDER (Gastrointestinal disorders) | 0 | 1
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTRIC INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 1 | 3
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 3
GINGIVAL BLEEDING (Gastrointestinal disorders) | 2 | 0
GINGIVITIS (Gastrointestinal disorders) | 1 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 2
HAEMORRHOIDS (Gastrointestinal disorders) | 2 | 1
HIATUS HERNIA (Gastrointestinal disorders) | 2 | 2
HYPERCHLORHYDRIA (Gastrointestinal disorders) | 1 | 0
ILEITIS (Gastrointestinal disorders) | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 2
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 | 1
MELAENA (Gastrointestinal disorders) | 1 | 0
MESENTERIC ARTERY STENOSIS (Gastrointestinal disorders) | 0 | 1
MESENTERIC PANNICULITIS (Gastrointestinal disorders) | 0 | 1
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 3 | 0
ORAL LICHEN PLANUS (Gastrointestinal disorders) | 1 | 0
PANCREATIC FISTULA (Gastrointestinal disorders) | 1 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 1
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 2
RECTAL POLYP (Gastrointestinal disorders) | 2 | 0
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 1 | 2
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 2
CHANGE OF BOWEL HABIT (Gastrointestinal disorders) | 0 | 1
ENTEROCOLITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 1
GASTRIC MUCOSAL LESION (Gastrointestinal disorders) | 0 | 1
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
ADVERSE DRUG REACTION (General disorders) | 14 | 30
CATHETER SITE HAEMATOMA (General disorders) | 4 | 6
CATHETER SITE HAEMORRHAGE (General disorders) | 5 | 8
CATHETER SITE PAIN (General disorders) | 1 | 6
CATHETER SITE PHLEBITIS (General disorders) | 0 | 1
CATHETER SITE SWELLING (General disorders) | 1 | 0
CHEST DISCOMFORT (General disorders) | 2 | 5
CHEST PAIN (General disorders) | 8 | 15
DEATH (General disorders) | 2 | 1
FATIGUE (General disorders) | 1 | 14
HERNIA (General disorders) | 1 | 0
MALAISE (General disorders) | 0 | 2
MASS (General disorders) | 1 | 0
MICROLITHIASIS (General disorders) | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 17 | 40
OEDEMA PERIPHERAL (General disorders) | 1 | 4
Other (General disorders) | 13 | 20
PELVIC MASS (General disorders) | 0 | 1
PERIODONTITIS (General disorders) | 0 | 1
PYREXIA (General disorders) | 1 | 1
SUDDEN DEATH (General disorders) | 0 | 1
THROMBOSIS IN DEVICE (General disorders) | 0 | 3
VASCULAR COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 0 | 1
ASTHENIA (General disorders) | 0 | 4
DRUG INTOLERANCE (General disorders) | 0 | 1
THIRST (General disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 2
HEPATIC CYST (Hepatobiliary disorders) | 0 | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 | 1
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 1 | 0
LIVER DISORDER (Hepatobiliary disorders) | 1 | 0
NON-ALCOHOLIC STEATOHEPATITIS (Hepatobiliary disorders) | 0 | 1
CONTRAST MEDIA ALLERGY (Immune system disorders) | 2 | 3
DRUG HYPERSENSITIVITY (Immune system disorders) | 4 | 1
HYPERSENSITIVITY (Immune system disorders) | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 1
ACARODERMATITIS (Infections and infestations) | 0 | 1
APPENDICITIS (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 7
CANDIDIASIS (Infections and infestations) | 0 | 2
CATHETER SITE ABSCESS (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 1
CHLAMYDIAL INFECTION (Infections and infestations) | 1 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 2
DOUGLAS' ABSCESS (Infections and infestations) | 1 | 0
EAR INFECTION (Infections and infestations) | 0 | 3
ERYSIPELAS (Infections and infestations) | 1 | 1
FUNGAL INFECTION (Infections and infestations) | 0 | 1
FUNGAL OESOPHAGITIS (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 2 | 3
GINGIVAL INFECTION (Infections and infestations) | 0 | 1
HELICOBACTER INFECTION (Infections and infestations) | 0 | 1
INFLUENZA (Infections and infestations) | 2 | 5
KIDNEY INFECTION (Infections and infestations) | 1 | 0
LABYRINTHITIS (Infections and infestations) | 0 | 1
LOCALISED INFECTION (Infections and infestations) | 1 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 5
LUNG INFECTION (Infections and infestations) | 1 | 0
LYMPHANGITIS (Infections and infestations) | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 2 | 7
ORCHITIS (Infections and infestations) | 0 | 2
OSTEOMYELITIS (Infections and infestations) | 1 | 0
PARONYCHIA (Infections and infestations) | 0 | 1
PHARYNGITIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 3 | 7
PYELONEPHRITIS (Infections and infestations) | 0 | 2
RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 7
SEPSIS (Infections and infestations) | 0 | 4
SEPTIC SHOCK (Infections and infestations) | 0 | 1
SINUSITIS (Infections and infestations) | 1 | 2
TOOTH INFECTION (Infections and infestations) | 2 | 1
URINARY TRACT INFECTION (Infections and infestations) | 4 | 1
UROSEPSIS (Infections and infestations) | 0 | 1
VAGINAL INFECTION (Infections and infestations) | 0 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 3
VULVAL ABSCESS (Infections and infestations) | 0 | 1
HERPES ZOSTER (Infections and infestations) | 1 | 1
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 | 0
CYSTITIS (Infections and infestations) | 0 | 4
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 2
HELICOBACTER GASTRITIS (Infections and infestations) | 0 | 1
HERPES OPHTHALMIC (Infections and infestations) | 1 | 0
LYME DISEASE (Infections and infestations) | 0 | 1
ORAL INFECTION (Infections and infestations) | 0 | 1
OTITIS EXTERNA (Infections and infestations) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 4
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 4
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 1 | 2
ESCHAR (Injury, poisoning and procedural complications) | 1 | 0
EXPOSURE TO CHEMICAL POLLUTION (Injury, poisoning and procedural complications) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 5 | 6
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 1 | 0
HAND FRACTURE (Injury, poisoning and procedural complications) | 3 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 | 1
LIGAMENT INJURY (Injury, poisoning and procedural complications) | 1 | 0
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 1 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 3
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
MOUNTAIN SICKNESS ACUTE (Injury, poisoning and procedural complications) | 1 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1 | 0
NERVE ROOT INJURY LUMBAR (Injury, poisoning and procedural complications) | 0 | 1
POISONING (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 | 0
POST PROCEDURAL MYOCARDIAL INFARCTION (Injury, poisoning and procedural complications) | 1 | 6
POSTOPERATIVE FEVER (Injury, poisoning and procedural complications) | 0 | 1
PROCEDURAL HEADACHE (Injury, poisoning and procedural complications) | 0 | 3
PROCEDURAL HYPERTENSION (Injury, poisoning and procedural complications) | 0 | 1
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 3 | 0
PROCEDURAL NAUSEA (Injury, poisoning and procedural complications) | 1 | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 3
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 2
SCIATIC NERVE INJURY (Injury, poisoning and procedural complications) | 0 | 1
SPINAL CORD INJURY (Injury, poisoning and procedural complications) | 0 | 2
SYNOVIAL RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 1
WOUND (Injury, poisoning and procedural complications) | 0 | 1
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
LIMB CRUSHING INJURY (Injury, poisoning and procedural complications) | 1 | 0
INJURY (Injury, poisoning and procedural complications) | 0 | 2
LACERATION (Injury, poisoning and procedural complications) | 0 | 4
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
CONFUSION POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 | 1
CONTRAST MEDIA ALLERGY (Injury, poisoning and procedural complications) | 1 | 1
EPICONDYLITIS (Injury, poisoning and procedural complications) | 0 | 1
EXPOSURE TO TOXIC AGENT (Injury, poisoning and procedural complications) | 0 | 1
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 0 | 6
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
TRAUMATIC ULCER (Injury, poisoning and procedural complications) | 0 | 1
ANGIOGRAM (Investigations) | 1 | 0
ANGIOTENSIN CONVERTING ENZYME INCREASED (Investigations) | 0 | 1
ARTERIOGRAM CORONARY (Investigations) | 1 | 1
BIOPSY PROSTATE (Investigations) | 0 | 1
BLOOD CHOLESTEROL INCREASED (Investigations) | 2 | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 2 | 5
BLOOD CREATINE PHOSPHOKINASE MB INCREASED (Investigations) | 4 | 5
BLOOD CREATININE INCREASED (Investigations) | 0 | 1
BLOOD GLUCOSE FLUCTUATION (Investigations) | 0 | 1
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 0
BLOOD PRESSURE INCREASED (Investigations) | 2 | 2
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1 | 0
BLOOD URINE PRESENT (Investigations) | 0 | 1
CARDIAC ENZYMES INCREASED (Investigations) | 35 | 74
CARDIAC STRESS TEST ABNORMAL (Investigations) | 5 | 6
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 0 | 2
ELECTROCARDIOGRAM ST SEGMENT ABNORMAL (Investigations) | 1 | 1
ELECTROCARDIOGRAM ST SEGMENT DEPRESSION (Investigations) | 2 | 2
ELECTROCARDIOGRAM ST SEGMENT ELEVATION (Investigations) | 0 | 2
EXERCISE TEST ABNORMAL (Investigations) | 1 | 2
GLYCOSYLATED HAEMOGLOBIN INCREASED (Investigations) | 1 | 0
HEART RATE INCREASED (Investigations) | 0 | 1
HEPATIC ENZYME INCREASED (Investigations) | 2 | 0
HIGH DENSITY LIPOPROTEIN DECREASED (Investigations) | 0 | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 2
TROPONIN I INCREASED (Investigations) | 12 | 30
TROPONIN INCREASED (Investigations) | 35 | 73
TROPONIN T INCREASED (Investigations) | 11 | 13
WEIGHT DECREASED (Investigations) | 0 | 1
BLOOD GLUCOSE ABNORMAL (Investigations) | 0 | 3
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1
HEART RATE DECREASED (Investigations) | 0 | 2
LOW DENSITY LIPOPROTEIN INCREASED (Investigations) | 0 | 3
STOOL ANALYSIS ABNORMAL (Investigations) | 0 | 1
TRANSAMINASES INCREASED (Investigations) | 0 | 1
WEIGHT INCREASED (Investigations) | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 | 5
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 | 3
GOUT (Metabolism and nutrition disorders) | 1 | 4
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 3
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
LIPID METABOLISM DISORDER (Metabolism and nutrition disorders) | 0 | 2
OBESITY (Metabolism and nutrition disorders) | 1 | 1
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 | 3
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 | 2
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERHOMOCYSTEINAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 8
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 8
DUPUYTREN'S CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 2
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 3
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 6
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 9
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 6
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 | 14
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 | 0
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PLANTAR FASCIITIS (Musculoskeletal and connective tissue disorders) | 2 | 1
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 0 | 1
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
TENOSYNOVITIS STENOSANS (Musculoskeletal and connective tissue disorders) | 1 | 0
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 2 | 3
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 | 1
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 | 2
SENSATION OF HEAVINESS (Musculoskeletal and connective tissue disorders) | 0 | 1
SJOGREN'S SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
BENIGN SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLON NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GASTROINTESTINAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
GASTROOESOPHAGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
GLIOBLASTOMA MULTIFORME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SMALL INTESTINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SMALL INTESTINE CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SWEAT GLAND TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SCROTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LEUKAEMIA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
AMNESIA (Nervous system disorders) | 0 | 1
APHASIA (Nervous system disorders) | 1 | 0
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 2 | 3
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 | 4
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 7 | 12
DIZZINESS POSTURAL (Nervous system disorders) | 0 | 5
DYSARTHRIA (Nervous system disorders) | 0 | 1
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 2 | 6
HYDROCEPHALUS (Nervous system disorders) | 1 | 0
HYPOKINESIA (Nervous system disorders) | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 2
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 3
PARAESTHESIA (Nervous system disorders) | 1 | 1
PARKINSON'S DISEASE (Nervous system disorders) | 0 | 1
PARKINSONISM (Nervous system disorders) | 0 | 1
POLYNEUROPATHY (Nervous system disorders) | 1 | 0
PRESYNCOPE (Nervous system disorders) | 2 | 2
SCIATICA (Nervous system disorders) | 1 | 1
SENSORY DISTURBANCE (Nervous system disorders) | 1 | 0
SENSORY LOSS (Nervous system disorders) | 2 | 0
SYNCOPE (Nervous system disorders) | 5 | 7
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 4 | 2
VIITH NERVE PARALYSIS (Nervous system disorders) | 0 | 1
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 0 | 1
LETHARGY (Nervous system disorders) | 0 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 1
EPILEPSY (Nervous system disorders) | 0 | 1
CLONIC CONVULSION (Nervous system disorders) | 0 | 1
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 1
MIGRAINE (Nervous system disorders) | 0 | 2
TREMOR (Nervous system disorders) | 0 | 1
ANXIETY (Psychiatric disorders) | 2 | 4
DEPRESSED MOOD (Psychiatric disorders) | 1 | 3
DEPRESSION (Psychiatric disorders) | 6 | 4
INSOMNIA (Psychiatric disorders) | 1 | 1
LIBIDO DECREASED (Psychiatric disorders) | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 2
MENTAL DISORDER (Psychiatric disorders) | 0 | 3
POST-TRAUMATIC STRESS DISORDER (Psychiatric disorders) | 0 | 1
PANIC ATTACK (Psychiatric disorders) | 0 | 1
SLEEP DISORDER (Psychiatric disorders) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 1 | 3
HYPERTONIC BLADDER (Renal and urinary disorders) | 1 | 0
RENAL COLIC (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0
RENAL PAIN (Renal and urinary disorders) | 0 | 1
URETHRAL STENOSIS (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 1
URINARY TRACT DISORDER (Renal and urinary disorders) | 0 | 2
VESICAL FISTULA (Renal and urinary disorders) | 1 | 0
CALCULUS URINARY (Renal and urinary disorders) | 0 | 1
POLLAKIURIA (Renal and urinary disorders) | 0 | 2
DYSURIA (Renal and urinary disorders) | 0 | 1
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 1 | 0
URETHRAL HAEMORRHAGE (Renal and urinary disorders) | 0 | 1
NOCTURIA (Renal and urinary disorders) | 0 | 1
RENAL ANEURYSM (Renal and urinary disorders) | 0 | 1
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 0 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 2 | 2
PROSTATISM (Reproductive system and breast disorders) | 0 | 1
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 | 3
SCROTAL PAIN (Reproductive system and breast disorders) | 0 | 1
BALANITIS (Reproductive system and breast disorders) | 0 | 1
PROSTATITIS (Reproductive system and breast disorders) | 0 | 1
CYSTOCELE (Reproductive system and breast disorders) | 0 | 1
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 | 2
PELVIC PAIN (Reproductive system and breast disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 9 | 12
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 11 | 20
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 10
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 | 6
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 4 | 0
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 2
RHINITIS ATROPHIC (Respiratory, thoracic and mediastinal disorders) | 0 | 1
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
VOCAL CORD LEUKOPLAKIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ALLERGIC COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
IDIOPATHIC PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PAINFUL RESPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 2
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 2 | 0
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 2 | 4
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 2 | 1
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 2
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0
BLISTER (Skin and subcutaneous tissue disorders) | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 3
DERMAL CYST (Skin and subcutaneous tissue disorders) | 1 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 2
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 1
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 0 | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 2
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 1
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 0 | 1
ELECTIVE PROCEDURE (Surgical and medical procedures) | 1 | 0
INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 1 | 0
SHOULDER OPERATION (Surgical and medical procedures) | 0 | 1
SPINAL LAMINECTOMY (Surgical and medical procedures) | 1 | 0
TOOTH EXTRACTION (Surgical and medical procedures) | 1 | 1
AORTIC ANEURYSM (Vascular disorders) | 2 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 1 | 1
HAEMATOMA (Vascular disorders) | 3 | 1
HYPERTENSION (Vascular disorders) | 8 | 21
HYPERTENSIVE CRISIS (Vascular disorders) | 4 | 1
HYPOTENSION (Vascular disorders) | 1 | 5
INTERMITTENT CLAUDICATION (Vascular disorders) | 1 | 3
ISCHAEMIA (Vascular disorders) | 0 | 1
PERIPHERAL COLDNESS (Vascular disorders) | 1 | 2
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 | 3
PHLEBITIS (Vascular disorders) | 1 | 0
TEMPORAL ARTERITIS (Vascular disorders) | 0 | 1
VARICOSE VEIN (Vascular disorders) | 0 | 1
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 0 | 1
AORTIC DILATATION (Vascular disorders) | 0 | 1
AORTIC STENOSIS (Vascular disorders) | 0 | 1
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 0 | 2
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 4
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 3
RAYNAUD'S PHENOMENON (Vascular disorders) | 0 | 1
CEREBRAL HAEMATOMA (Nervous system disorders) | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CATHETER SITE HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less